CLINICAL TRIAL: NCT06064318
Title: Prevalence and Incidence of Multiple Revisions Following Knee Arthroplasty in Denmark 1998-2021: A Nationwide Population-based Study
Acronym: EMKAR ONE
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Julius Tetens Hald, Dr., Rigshospitalet, Denmark
Other Study IDs: 08062023
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Knee Replacement; Knee Replacement Revision
MeSH Terms: interventions — Second-Look Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary cohort: All patients with a primary knee arthroplasty performed in Denmark between Jan 1st 1998 and 31st December 2021.
- Revision cohort: All patients with a revision knee arthroplasty performed in Denmark between Jan 1st 1998 and 31st December 2021
  Interventions: Procedure: Revision

INTERVENTIONS:
Procedure: Revision — Any type of knee revision, excluding knee arthrodesis and femur amputation
  Groups: Revision cohort

SUMMARY:
The purpose of this study is to investigate the incidence and prevalence rates of multiply revised knee arthroplasty patients in Denmark from 1998-2021.

ELIGIBILITY:
Inclusion Criteria:

* Danish Resident
* all ages
* must have had primary knee arthroplasty procedure performed in Denmark between 1998-2021

Exclusion Criteria:

* Missing key variables (patient ID, date of surgery, procedure-code, laterality of procedure)
* Duplicates
* Non-relevant procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Danish residents who received a primary knee arthroplasty in Denmark between 1998-2021.
Sampling Method: Non-Probability Sample
Enrollment: 161384 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of major n-grade revisions | 23 years
  standardized prevalence of major n-grade revisions
Incidence of major n-grade revisions | 23 years
  standardized incidence of major n-grade revisions
Prevalence of all n-grade revisions | 23 years
  standardized prevalence of all n-grade revisions
Incidence of all n-grade revisions | 23 years
  standardized incidence of all n-grade revisions

SECONDARY OUTCOMES:
Incidence of major and all n-grade revisions stratified by sex and age | 23 years
  Calculation of incidence for major and for all n-grade revisions stratified by sex and by age (groups, sex: male/female, age: 18-49/50-69/70-99)
Prevalence of major and all n-grade revisions stratified by sex and age | 23 years
  Calculation of prevalence for major and for all n-grade revisions stratified by sex and by age (groups, sex: male/female, age: 18-49/50-69/70-99)
Prevalence of major and all n-grade revisions for patients with their total sum of revisions | 23 Years
  Calculation of standardized prevalence for patients receiving major or all type of n-grade revision, where the ordering of revisions are not knee specific but patient-specific

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is not available as the data is protected by GDPR regulations.

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT06064318/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT06064318/SAP_001.pdf